CLINICAL TRIAL: NCT02989909
Title: Clinical Evaluation of CATS Tonometer Prism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CATS Tonometer, LLC - CP-01
Record Dates: First submitted 2016-11-28; First posted 2016-12-12 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goldmann Tonometer (Active Comparator): Goldmann Tonometer prism will be used as a based line comparator for tolerance assessment versus the active test comparator CATS tonometer prism
  Interventions: Device: Goldmann tonometer prism
- CATS tonometer (Experimental): CATS tonometer prism being used as the test product to assess IOP measurement versus active comparator the Goldmann Tonometer prism
  Interventions: Device: CATS tonometer prism

INTERVENTIONS:
Device: CATS tonometer prism — demonstrate that not more than 5% of the paired differences between the reference tonometer (CATS prism) reading and the test tonometer (Goldmann prism) reading for each pressure range
  Arms: CATS tonometer
Device: Goldmann tonometer prism — demonstrate that not more than 5% of the paired differences between the reference tonometer (CATS prism) reading and the test tonometer (Goldmann prism) reading for each pressure range
  Arms: Goldmann Tonometer

SUMMARY:
Prospective, open-labeled, randomized, controlled, multicenter study at two clinical investigative sites in Tucson, Arizona. The subjects will undergo intraocular pressure measurement with the CATS tonometer prism and the Goldmann applanation tonometer prism (GAT).

Of the 200 eyes, at least 10 highly astigmatic eyes (>3 D of corneal astigmatism) each in the low, medium and high IOP ranges shall have the same clinical testing and analysis of results, with the analysis kept separate from that of the main group.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable)obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Male and female patients, at least 18 years of age

Exclusion Criteria:

* Subject has undergone ocular surgery within the last 3 months
* Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's heath at risk
* Pregnant or nursing women
* Subjects with only one functional eye
* Those with one eye having poor or eccentric fixation
* Eyes displaying an oval contact image
* Those with corneal scarring or who have had corneal surgery including corneal laser surgery
* Microphthalmos
* Buphthalmos
* Contact lens wearers
* Severe Dry eyes
* Lid squeezers - blepharospasm
* Nystagmus
* Keratoconus
* Any other corneal or conjunctival pathology or infection.
* Central corneal thickness greater than 0.600 mm or less than 0.500 mm (2 standard deviations about the human mean)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
All subjects will have CATS tonometer prism intraocular pressure readings compared to Goldmann tonometer prism readings in establishing effectiveness. | From date of randomization until 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Eye Consultants, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCafferty SJ, Tetrault K, McColgin A, Chue W, Levine J, Muller M. Modified Goldmann prism intraocular pressure measurement accuracy and correlation to corneal biomechanical metrics: multicentre randomised clinical trial. Br J Ophthalmol. 2019 Dec;103(12):1840-1844. doi: 10.1136/bjophthalmol-2018-313470. Epub 2019 Feb 22. PMID 30796054